CLINICAL TRIAL: NCT07161167
Title: Changes in Body Composition of Patients With Obesity Related Tumors and Their Impact on Clinical Outcomes: a Multicenter Prospective Cohort Study
Status: Not yet recruiting | Type: Observational
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: obesity-related cancer & BC
Record Dates: First submitted 2025-07-21; First posted 2025-09-08 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-07

CONDITIONS: Obesity Rekated Cancer; Body Composition Changes; Survival; Mechanism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Over the past 20 years, China's obesity rates have surged, increasing cancer burden. Obesity links to 13 cancers via metabolic effects of visceral fat and insulin resistance, while sarcopenic obesity (BMI-independent) may worsen outcomes. Traditional BMI lacks precision; advanced methods (e.g., BIA/CT) are needed. Existing studies show inconsistent results, possibly due to heterogeneity. This multicenter prospective cohort study uses imaging to assess body composition changes (fat/muscle) in obesity-related tumors and their impact on survival, recurrence, and quality of life, and explore the underlying mechanism.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years, regardless of gender.
2. Histologically or cytologically confirmed obesity-associated malignant tumors (e.g., breast cancer, colorectal cancer, gastric cancer, lung cancer, or thyroid cancer) with planned treatment after diagnosis (any treatment modality permitted).
3. No prior chemotherapy, radiotherapy, biologic therapy, immunotherapy, or other antitumor treatments for malignancy.

Exclusion Criteria:

1. Patients with concurrent non-obesity-related malignancies.
2. History of prior malignancy (except completely cured carcinoma in situ of the cervix, basal cell carcinoma, or squamous cell carcinoma of the skin).
3. Patients with concurrent multiorgan dysfunction syndrome, autoimmune diseases, infectious diseases, neurological disorders, or psychiatric disorders.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study participants will be enrolled if they are under clinical care in oncology-related departments
Sampling Method: Non-Probability Sample
Enrollment: 6743 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2030-09-30 (Estimated); Study Completion 2030-09-30 (Estimated)

PRIMARY OUTCOMES:
Overall survival | From date of diagnosis until the date of death from any cause, assessed up to 10 years
  The time from the start of follow-up to death (for any reason).

SECONDARY OUTCOMES:
Progression-free survival after diagnosis | From date of diagnosis until the date of first documented progression , assessed up to 10 years
Time of recurrence and/or distant metastasis after diagnosis | From date of diagnosis until the date of first documented recurrence and/or distant metastasis, whichever came first, assessed up to 10 years

CONTACTS AND LOCATIONS:
Locations (1):
- Peking union medical college hospital, Beijing, Beijing Municipality, China